CLINICAL TRIAL: NCT06295367
Title: Effectiveness of Out-of-Pocket Cost COMmunication and Financial Navigation (CostCOM) in Cancer Patients
Brief Title: Cost Communication and Financial Navigation in Cancer Patients (COSTCOM)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: EAQ222CD; NCI-2023-09944 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAQ222CD (Other: ECOG-ACRIN Cancer Research Group); ECOG-ACRIN-EAQ222CD (Other: DCP); EAQ222CD (Other: CTEP); R01CA272680 (NIH); UG1CA189828 (NIH)
Record Dates: First submitted 2024-02-14; First posted 2024-03-06 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Malignant Solid Neoplasm
MeSH Terms: interventions — Practice Guidelines as Topic; Standard of Care; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ARM A (Enhanced usual care) (Active Comparator): Patients receive PAF brochure describing financial navigation services.
  Interventions: Other: Best Practice; Other: Survey Administration
- ARM B (CostCOM) (Experimental): Patients receive usual financial care per practice standard of care and CostCOM financial counseling sessions over 1 hour within 30 days after enrollment and at 3, 6 and 12 months.
  Interventions: Other: Best Practice; Other: Financial Navigation; Other: Survey Administration
- Non-patient participants: (interview) (Experimental): Non-patient participants complete surveys and participant in 1 on 1 in depth semi-structured interview over 20-30 minutes at 15-39 months after first patient enrollment.
  Interventions: Other: Interview; Other: Survey Administration

INTERVENTIONS:
Other: Best Practice — Receive PAF brochure describing financial navigation services
  Other Names: standard of care; standard therapy
  Arms: ARM A (Enhanced usual care); ARM B (CostCOM)
Other: Financial Navigation — Receive CostCOM financial counseling
  Other Names: Financial Navigation Program
  Arms: ARM B (CostCOM)
Other: Interview — Participate in a 1 on 1 in-depth interview
  Arms: Non-patient participants: (interview)
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial evaluates the effect of Cost Communication and Financial Navigation (CostCOM) intervention on adherence to care and financial burden in cancer patients. Many cancer patients experience financial hardship due to high medical out of pocket costs (OOPC), changes in employment, income and insurance. Financial hardship can lead to a delay or a stop in cancer care, and is linked to poor quality of life. Financial navigation programs, such as CostCOM, provide financial counseling, education and connections to appropriate resources to reduce financial barriers to healthcare and minimize financial stress and burden. CostCOM may improve adherence to care and decrease financial burden in patients with cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare patient-reported cost-related cancer care non-adherence at 12 months after completion of baseline survey between the enhanced usual care (EUC) and CostCOM study arms.

SECONDARY OBJECTIVES:

I. To compare patient-reported material financial hardship at 12 months after completion of baseline survey between the EUC and CostCOM study arms.

II. To compare patient-reported financial worry at 12 months after completion of baseline survey between the EUC and CostCOM study arms.

III. To compare patient-reported quality of life at 12 months after completion of baseline survey between the EUC and CostCOM study arms.

IV. To compare patient satisfaction with care at 12 months after completion of baseline survey between the EUC and CostCOM study arms.

EXPLORATORY OBJECTIVES:

I. To describe CostCOM (Arm B) patients and their provider experience with various implementation outcomes.

II. To assess accuracy of out-of-pocket estimates communicated with the CostCOM (Arm B) patients at part of the intervention with their reported actual out-of-pocket cost.

III. To compare neighborhood characteristics of patient participants versus (vs.) practice patient population.

IV. To assess patients' satisfaction with CostCOM in patients with Arm B. V. To assess patients' receipt of financial navigation via internal practice or external resources.

VI. To evaluate longitudinal changes in cost-related cancer care non-adherence, material hardship, financial worry, quality of life and satisfaction with care.

OUTLINE:

Non-patient participants: Participants complete surveys and participant in 1 on 1 in depth semi-structured interview over 20-30 minutes at 15-39 months after first patient enrollment.

Patients are randomized to 1 of 2 arms.

ARM A: Patients receive Patient Advocate Foundation (PAF) brochure describing financial navigation services.

ARM B: Patients receive usual financial care per practice standard of care and CostCOM financial counseling sessions over 1 hour within 30 days after enrollment and at 3, 6 and 12 months.

Patients are followed up within 12 months of study intervention completion.

ELIGIBILITY:
Inclusion Criteria:

* NON-PATIENTS PARTICIPANTS: Participant must speak English
* NON-PATIENTS PARTICIPANTS: Participant must be employed at National Cancer Institute Community Oncology Research Program (NCORP) site for at least six months
* NON-PATIENTS PARTICIPANTS: Participant must be able to provide informed consent to participate in this study
* NON-PATIENTS PARTICIPANTS: Participant must be one of the following:

  * A study coordinator with a role involving use of CostCOM intervention price transparency and financial navigation platform
  * A practice oncology provider (i.e., physician or mid-level), or
  * A practice financial counselor, social workers, financial navigators, or pharmacist who have provided care or been in contact (in the last 3 months) to a patient who was assigned to the CostCOM arm, and who completed the at least 6 month study follow-up
* PATIENT ELIGIBILITY CRITERIA FOR STEP 0 (OPEN SCREENING REGISTRATION): Patient must be ≥ 18 years of age
* PATIENT ELIGIBILITY CRITERIA FOR STEP 0 (OPEN SCREENING REGISTRATION): Patient must be fluent in written and spoken English OR patient must be fluent in written and spoken Spanish
* PATIENT ELIGIBILITY CRITERIA FOR STEP 0 (OPEN SCREENING REGISTRATION): Patient must be within 120 days of a new diagnosis of any solid cancer of any stage at the time of Step 0
* PATIENT ELIGIBILITY CRITERIA FOR STEP 0 (OPEN SCREENING REGISTRATION): Patient must have had their first medical oncology visit at the time of Step 0
* PATIENT ELIGIBILITY CRITERIA FOR STEP 0 (OPEN SCREENING REGISTRATION): Patient must have initiated oral or intravenous (IV) cancer systemic therapy or have received a prescription order with stated intent to initiate within 30 days following Step 0 consent
* PATIENT ELIGIBILITY CRITERIA FOR STEP 0 (OPEN SCREENING REGISTRATION): Patients must not have indolent cancer undergoing observation alone (i.e., active surveillance)
* PATIENT ELIGIBILITY CRITERIA FOR STEP 0 (OPEN SCREENING REGISTRATION): Patients must not be receiving palliative or hospice care alone
* PATIENT ELIGIBILITY CRITERIA FOR STEP 0 (OPEN SCREENING REGISTRATION): Patient must not be undergoing curative surgery alone or radiation therapy alone. (Must be receiving systemic therapy), unless they are receiving systemic therapy
* PATIENT ELIGIBILITY CRITERIA FOR STEP 0 (OPEN SCREENING REGISTRATION): Patient must confirm that they intend to receive their care or monitoring at one of the participating NCORP practices
* PATIENT ELIGIBILITY CRITERIA FOR STEP 0 (OPEN SCREENING REGISTRATION): Patient must have the ability to understand and the willingness to sign a written informed consent document.

  * Patients with impaired decision-making capacity (IDMC) who have a legally authorized representative (LAR) or caregiver and/or family member available are not eligible
* PATIENT ELIGIBILITY CRITERIA FOR STEP 0 (OPEN SCREENING REGISTRATION): Patient must not have an Eastern Cooperative Oncology Group (ECOG) performance status ≥ 3, OR

  * Patient must not be deemed medically unable to participate in the study by the study investigators or an oncology clinician (i.e., referral to hospice)
* PATIENT ELIGIBILITY CRITERIA FOR STEP 0 (OPEN SCREENING REGISTRATION): Patient must not be enrolled in treatment clinical trials where cancer systemic therapy is provided at no cost to the patient
* PATIENT ELIGIBILITY CRITERIA FOR STEP 0 (OPEN SCREENING REGISTRATION): Patient must not be enrolled in EAQ221CD or S1912CD given financial navigation is offered as part of these two trials.

  * NOTE: If S1912CD is activated in a participating practice, S1912CD should be offered first to patients with metastatic cancer meeting eligibility criteria for S1912CD. Only if a patient is not eligible or not interested in participating in S1912CD, the EAQ222CD can be offered. For early stage cancer, EAQ222CD can be offered first given S1912CD does not enroll patients with early stage cancer
* PATIENT ELIGIBILITY CRITERIA FOR STEP 0 (OPEN SCREENING REGISTRATION): Patient must not be enrolled in other clinical trials where OOPC communication or financial navigation (i.e., professional guidance to identify financial assistance programs to alleviate cost of care) is being offered as part of the trial

  * NOTE: If a trial is offering financial counseling alone without financial navigation patients are allowed to co-enroll
  * NOTE: Gift cards for survey completion, or parking passes are not considered financial navigation
* PATIENT ELIGIBILITY CRITERIA FOR STEP 1 (OPEN RANDOMIZATION): Patient must meet all the eligibility criteria for step 0
* PATIENT ELIGIBILITY CRITERIA FOR STEP 1 (OPEN RANDOMIZATION): Patient must have signed a written informed consent form
* PATIENT ELIGIBILITY CRITERIA FOR STEP 1 (OPEN RANDOMIZATION): Patient must have a completed baseline survey in ECOG American College of Radiology Imaging Network Systems for Easy Entry of Patient Reported Outcomes (EASEE-PRO) within 30 days of the date of OPEN registration and consent (step 0)
* PATIENT ELIGIBILITY CRITERIA FOR STEP 1 (OPEN RANDOMIZATION): Patients must have initiated their cancer treatment (i.e., IV or oral systemic therapy) either before or within 30 days of the date of OPEN registration and consent (step 0)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 760 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Cost-related cancer care non-adherence | 12 months
  Cost-related cancer care non-adherence is defined as a positive response to any of the following due to costs: Delayed, forewent, stopped, or changed prescribed cancer medication; or delayed, forewent, or refused recommended cancer tests, or cancer office visits. Will be calculated as a report of non-adherence at any point up through the 12mo follow-up survey.

SECONDARY OUTCOMES:
Rate of Material Financial Hardship | at 12 months
  Rate of material hardship at each time point is a binary (yes/no) composite measure defined as a positive response to any of the following: (1) home sale, refinance or move to affordable rental, (2) loans, (3) reaching credit limits, and (4) bankruptcy because of your cancer care, or its treatment (adapted from Medical Expenditure Panel Survey).Material hardship at 12 months is measured as report of material hardship at any of the 3, 6 and 12 follow-ups.
Patient-reported financial worry | At baseline and at 3, 6 and 12 months
  Measured by 12-item Comprehensive Score for Financial Toxicity (de Souza COST measure). Composite Scores range between 0-44 with higher the scores reflecting better the Financial Well-Being. Item 12 , an unscored summary item, will be used separately as a single item measure of financial worry. Mean score and changes in mean scores from baseline at each time point between the arms will be compared using two-sample t-tests.
Patient-reported Quality of life - mental and physical health | At baseline and at 3, 6 and 12 months
  Measured using the 10-item Patient-Reported Outcomes Measurement Information System (PROMIS-10) version 1.2 Global Health. A T-score will be calculated for each of the global mental health and global physical health sections with a higher PROMIS T-score representing more of the concept being measured (mental/physical health). T-scores for the general population have a mean of 50 and a standard deviation (SD) of 10.Thus, a person who has T- scores of 60 for the Global Physical Health or Global Mental Health scales is one standard deviation better (more healthy) than the general population Mean score and changes in mean scores from baseline at each time point between the arms will be compared using two-sample t-tests.
Patient-reported satisfaction with care at 12 months | At baseline and at 3, 6 and 12 months
  Satisfaction with the care will be measured using Consumer Assessment of Healthcare Providers and Systems (CAHPS) Cancer Care Survey questions. Composite items are rated on a scale of 0 to 10, with 0 being the worst and 10 being the best. Mean score and changes in mean scores from baseline at each time point between the arms will be compared using two-sample t-tests.

OTHER OUTCOMES:
Out of pocket cost (OOPC) accuracy | At 3, 6 and 12 months
  Mean absolute difference between OOPC estimates for the first cycle of therapy (as estimated by TailorMed Medical Incorporated) and the actual billed out of pocket (OOP) costs (as reported by patients based on their co-pays or medical bills).
Proportion of study patient participants that are of minority racial/ethnic background, and with public insurance will be measured and compared with that of practice patient population. | Up to 12 months
  Proportion of patients with specific characteristics, including racial, ethnic, payer mix, and neighborhood deprivation indices. Proportions will be compared between study participants and practice patient population.
Patient reported satisfaction with intervention | 39 months after enrollment of first study participant
  Qualitative interviews utilizing the Reach, Effectiveness, Adoption, Implementation and Maintenance (RE-AIM) framework was used to guide the evaluation questions and examine the effectiveness of the intervention and implementation outcomes.
  Participants describe their experience with various components of the CostCOM intervention: price transparency, financial navigation, and financial counseling, barriers and facilitators to participation, and feedback on what they liked and disliked about CostCOM, how it impacted their care, satisfaction with care, and what they would change to make it more helpful or engaging. The outcome measures are the proportion of subjects in the top 10 categories identified (5 for each like and dislike)
Receipt of financial navigation via internal practice or external resources | 12 months
  Proportion of subjects receiving (at least 1 session) of financial navigation via study intervention, internal practice, or external resources.
  Receipt of financial counseling or financial assistance will be documented via treating clinic as extracted from medical records and intervention participants via reports from TailorMed Medical Incorporated
Evaluate longitudinal changes in Cost-related cancer care non-adherence, material hardship, financial worry, quality of life and satisfaction with care | At baseline and at 3, 6 and 12 months
  Cost-related cancer care outcomes of non-adherence, material hardship, financial worry, quality of life and satisfaction with care (reported above) are included in a Regression Model (GEE)
longitudinal changes in cost-related cancer care non-adherence | At baseline, 3, 6 and 12 months
  The effect of time (unitless Betas (slope)) will be estimated using a regression model (stage-stratified GEE analyses) for the Cost-related Outcomes non-adherence, material hardship, financial worry, quality of life, and satisfaction with care Regression intervention parameter (COSTCOM v EUC) will use EUC as the reference category.
  Cost-related cancer care non-adherence is defined as a positive response to any of the following due to costs: Delayed, forewent, stopped, or changed prescribed cancer medication; or delayed, forewent, or refused recommended cancer tests, or cancer office visits
longitudinal changes in cost-related cancer care material hardship | At baseline, 3, 6 and 12 months
  The effect of time (unitless Betas (slope)) will be estimated using a regression model (stage-stratified GEE analyses) for the Cost-related Outcomes non-adherence, material hardship, financial worry, quality of life, and satisfaction with care Regression intervention parameter (COSTCOM v EUC) will use EUC as the reference category.
  Material hardship is a binary (yes/no) composite measure defined as a positive response to any of the following: (1) home sale, refinance or move to affordable rental, (2) loans, (3) reaching credit limits, and (4) bankruptcy because of your cancer care, or its treatment (adapted from Medical Expenditure Panel Survey).
longitudinal changes in cost-related cancer care financial worry | At baseline, 3, 6 and 12 months
  The effect of time (unitless Betas (slope)) will be estimated using a regression model (stage-stratified GEE analyses) for the Cost-related Outcomes non-adherence, material hardship, financial worry, quality of life, and satisfaction with care Regression intervention parameter (COSTCOM v EUC) will use EUC as the reference category.
  Financial Worry measured by the 12-item Comprehensive Score for Financial Toxicity (de Souza COST measure). Composite Scores range between 0-44 with higher the scores reflecting better the Financial Well-Being. Item 12 , an unscored summary item, will be used separately as a single item measure of financial worry. Mean score and changes in mean scores from baseline at each time point between the arms will be compared using two-sample t-tests.
longitudinal changes in cost-related cancer care quality of life | At baseline, 3, 6 and 12 months
  The effect of time (unitless Betas (slope)) will be estimated using a regression model (stage-stratified GEE analyses) for the Cost-related Outcomes non-adherence, material hardship, financial worry, quality of life, and satisfaction with care Regression intervention parameter (COSTCOM v EUC) will use EUC as the reference category.
  Quality of life is measured using the 10-item Patient-Reported Outcomes Measurement Information System (PROMIS-10) ver 1.2 Global Health. A T-score will be calculated for each global mental health and global physical health sections with a higher PROMIS T-score representing more of the concept being measured (mental/physical health). T-scores for the general population have a mean of 50 and a standard deviation (SD) of 10.Thus, a person who has T- scores of 60 for the Global Physical Health or Global Mental Health scales is one standard deviation better (more healthy) than the general population Mean score and changes in mean scores from base
longitudinal changes in cost-related cancer care satisfaction with care | At baseline, 3, 6 and 12 months
  The effect of time (unitless Betas (slope)) will be estimated using a regression model (stage-stratified GEE analyses) for the Cost-related Outcome Satisfaction with care Regression intervention parameter (COSTCOM v EUC) will use EUC as the reference category.
  Satisfaction with the care is measured using the Consumer Assessment of Healthcare Providers and Systems (CAHPS) Cancer Care Survey questions. Composite items are rated on a scale of 0 to 10, with 0 being the worst and 10 being the best.

CONTACTS AND LOCATIONS:
Overall Officials: Gelareh Sadigh, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (181):
- United States (174):
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CARTI Cancer Center, Little Rock, Arkansas
  - Contra Costa Regional Medical Center, Martinez, California
  - BASS Medical Group - Lennon, Walnut Creek, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Rocky Mountain Cancer Centers - Centennial, Centennial, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Rocky Mountain Cancer Centers - Swedish, Englewood, Colorado
  - The Melanoma and Skin Cancer Institute, Englewood, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Diagnostic Radiology Services LLC, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Straub Medical Center - Kahului Clinic, Kahului, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - The Queen's Medical Center - West Oahu, ‘Ewa Beach, Hawaii
  - Saint Anthony's Health, Alton, Illinois
  - Saint Mary's Hospital, Centralia, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Mercy Health - Paducah Medical Oncology and Hematology, Paducah, Kentucky
  - Bronson Battle Creek, Battle Creek, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Ascension Borgess Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Lake Regional Hospital, Osage Beach, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Cone Health Cancer Center at Asheboro, Asheboro, North Carolina
  - Randolph Health Cancer Center, Asheboro, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Cone Health Cancer Center at Drawbridge Parkway, Greensboro, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Central Ohio Breast and Endocrine Surgery, Gahanna, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Zangmeister Center Grove City, Grove City, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Memorial Hospital, Marysville, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Mount Carmel New Albany Surgical Hospital, New Albany, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Mercy Health Perrysburg Cancer Center, Perrysburg, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Mercy Health - Saint Vincent Hospital, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Mercy Health Sylvania Radiation Oncology Center, Toledo, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Clinton Memorial Hospital/Foster J Boyd Regional Cancer Center, Wilmington, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Medical Oncology-Selinsgrove, Selinsgrove, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - Bon Secours Westchester Emergency Center, Midlothian, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Bon Secours Richmond Community Hospital, Richmond, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - Bon Secours Cancer Institute at Reynolds Crossing, Richmond, Virginia
  - Jefferson Healthcare, Port Townsend, Washington
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Ascension Saint Elizabeth Hospital, Appleton, Wisconsin
  - ThedaCare Cancer Care - Berlin, Berlin, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Elmbrook Campus, Brookfield, Wisconsin
  - Ascension Calumet Hospital, Chilton, Wisconsin
  - Ascension Saint Francis - Reiman Cancer Center, Franklin, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Franklin, Franklin, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Ascension Columbia Saint Mary's Hospital Ozaukee, Mequon, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Saint Joseph Campus, Milwaukee, Wisconsin
  - Ascension Columbia Saint Mary's Hospital - Milwaukee, Milwaukee, Wisconsin
  - Ascension Saint Francis Hospital, Milwaukee, Wisconsin
  - ThedaCare Regional Medical Center - Neenah, Neenah, Wisconsin
  - ThedaCare Cancer Care - New London, New London, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Ascension Mercy Hospital, Oshkosh, Wisconsin
  - ThedaCare Cancer Care - Oshkosh, Oshkosh, Wisconsin
  - Ascension All Saints Hospital, Racine, Wisconsin
  - ThedaCare Cancer Care - Shawano, Shawano, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - ThedaCare Cancer Care - Waupaca, Waupaca, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Ascension Medical Group Southeast Wisconsin - Mayfair Road, Wauwatosa, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
- Puerto Rico (7):
  - Cancer Center-Metro Medical Center Bayamon, Bayamón
  - Puerto Rico Hematology Oncology Group, Bayamón
  - Doctors Cancer Center, Manatí
  - San Juan Community Oncology Group, San Juan
  - Centro Comprensivo de Cancer de UPR, San Juan
  - PROncology, San Juan
  - San Juan City Hospital, San Juan

REFERENCES:
- [Derived] Sadigh G, Duan F, Gareen IF, Hancock J, Sicks JD, Hawley S, Shankaran V, Torres M, Wagner LI, Carlos RC. Effectiveness of out-of-pocket cost COMmunication and financial navigation (CostCOM) in cancer patients: Study protocol for ECOG-ACRIN EAQ222CD. Contemp Clin Trials. 2025 Jun;153:107889. doi: 10.1016/j.cct.2025.107889. Epub 2025 Mar 25. PMID 40147544